CLINICAL TRIAL: NCT03882658
Title: Preoperative Serum Albumin and Duration of Intraoperative Hypotension on Postoperative Acute Kidney Injury: a Retrospective Cohort Analysis
Brief Title: Preoperative Serum Albumin and Duration of Intraoperative Hypotension on Postoperative Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, Principal Investigator, Peking University First Hospital
Other Study IDs: ALBHYTAKI
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury is one of major adverse postoperative complications. research about postoperative acute kidney injury conclude that low preoperative albumin and intraoperative hypotension is associated to postoperative acute kidney injury. However, due to ethic issue and nonlinear realtionship between these factors and postoperative acute kidney injury, the exact threshold of these two risk factors were not be able to identified. The research tried to locate the exact threshold with implementation of penalized splines by generalized additive model.

ELIGIBILITY:
Inclusion Criteria:

adult non-cardiac, non-obsteric, non- kidney elective surgery patients

Exclusion Criteria:

patients aged <18 y emergency surgeries without arterial blood pressure cardiac surgeries obstetric surgeries kidney surgeries under local infiltration or MAC first SBP <100 mmHg

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult non-cardiac, non-obsteric, non- kidney elective surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 37610 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
incidence and odds ratio of postoperative acute kidney injury | 30 days postoperatively in hospital
  incidence and odds ratio of postoperative acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhou, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- First hospital Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No